CLINICAL TRIAL: NCT03209856
Title: Vitamin D Supplementation in Vitamin Deficient Women Undergoing ICSI Cycles: Does it Affect the Fertility Outcome?
Brief Title: Vitamin D Supplementation in Vitamin Deficient Women Undergoing IVF Cycles: Does it Affect the Fertility Outcome?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Omran, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3645
Record Dates: First submitted 2017-07-04; First posted 2017-07-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Vitamin D; Calcitriol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D supplement (Experimental): This group will receive weekly oral 50000 international units of vitamin D supplement for 8 weeks before the start of ICSI cycle. In addition, the routine care will be given.
  Interventions: Drug: Vitamin D
- Routine care (No Intervention): This group will receive the routine care.

INTERVENTIONS:
Drug: Vitamin D — Vitamin D supplement will be given. Then, it will be maintained if pregnancy occurred
  Other Names: Calcitriol
  Arms: Vitamin D supplement

SUMMARY:
The aim of this study is to evaluate the effect of treatment of vitamin D deficiency (through vitamin D supplementation for 8 weeks before the start of In-vitro fertilization (IVF) on the success of IVF cycles.

DETAILED DESCRIPTION:
The study participants are vitamin D deficient females undergoing (intra-cytoplasmic sperm injection (ICSI) trial in the age of 20 to 35 years. Serum vitamin D will be assessed. Accordingly, if they are deficient in vitamin D, they will be eligible for the study.400 vitamin D deficient women will be randomly allocated to either one of two groups. The first group will receive vitamin D supplementation in addition to the routine care. The other group will receive the routine care only. The study will be conducted in the IVF unit of department of Obstetrics and Gynecology, Cairo University.

ELIGIBILITY:
Inclusion Criteria:

* Vitamin D deficient females undergoing first ICSI trial
* Age from 20 to 35 years

Exclusion Criteria:

* Women undergoing ICSI trials who are vitamin D sufficient

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | It will be calculated 1 year after enrollment of the first patient in the study
  This outcome will be calculated by a statistician

CONTACTS AND LOCATIONS:
Overall Officials: Eman Omran, M.D., Principal Investigator — Cairo University
Locations (1):
- Department of Obstetrics and Gynecology, Kasr Al-Ainy hospital, Cairo, Greater Cairo, Egypt